CLINICAL TRIAL: NCT05522348
Title: Stability of Two Different Designs of Patient Specific Osteosynthesis "One Piece VS Two Piece" For The Fixation of LeFort 1 Osteotomy in Maxillary Orthognathic Surgery A Randomized Clinical Trial
Brief Title: Stability of Two Designs of Patient Specific Osteosynthesis For Fixation of LeFort 1 Osteotomy in Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shady Medhat Sabet Shaker, Master's degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2021-10-24
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Dentofacial Deformities
Keywords: Computer guided orthognathic surgery; Splintless orthognathic surgery; Patient specific osteosynthesis; stability of le fort 1 osteotomy
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Intervention Model Description: randomized clinical trial parallel study and control groups equal randomization positive controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcome assessor will be blinded to the intervention, however the primary investigator will not be blinded as he performs the surgical procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stability of a two piece PSI deign in splintless maxillary orthognathic surgery (Experimental): A two piece fixation device will be used connecting the nasomaxillary and the zygomaticomaxillary buttresses on both sides
  Interventions: Procedure: Stability of a two piece PSI deign in splintless maxillary orthognathic surgery
- Stability of a one piece PSI deign in splintless maxillary orthognathic surgery (Active Comparator): A one piece fixation device will be used extending from one zygomaticomaxillary buttress to the nasomaxillary area then just below the anterior nasal spine then to the same buttresses on the other side
  Interventions: Procedure: Stability of a one piece PSI deign in splintless maxillary orthognathic surgery

INTERVENTIONS:
Procedure: Stability of a two piece PSI deign in splintless maxillary orthognathic surgery — two patient fitted custom made plates will be used for the fixation of the maxilla following le fort 1 osteotomy for the correction of the dentofacial deformity and the postoperative stability will be measured using postoperative xrays
  Arms: Stability of a two piece PSI deign in splintless maxillary orthognathic surgery
Procedure: Stability of a one piece PSI deign in splintless maxillary orthognathic surgery — one patient fitted custom made plate will be used for the fixation of the maxilla following le fort 1 osteotomy for the correction of the dentofacial deformity and the postoperative stability will be measured using postoperative xrays
  Arms: Stability of a one piece PSI deign in splintless maxillary orthognathic surgery

SUMMARY:
A comparison of the stability of two different designs of patient specific fixation devices for the performance of splintless computer guided le fort 1 osteotomy in orthognathic surgery workflow for the correction of a variety of dentofacial deformities

DETAILED DESCRIPTION:
• Intervention Group: -

Pre-Operative Virtual planning:

After CT examinations, further processing of the DICOM files (Digital Imaging and Communications in Medicine) will be performed using the specialized DICOM image processing software and reconstructed 3D models of the skull will be made. Stone models will be scanned using an optical scanner and stereolithographic files will be imported. Registration of the STL files with the skull model will create a composite model suitable for the construction of necessary devices. These 3D models will be used to design the custom-made cutting guides and fixation devices. The final STL files will be sent to the lab to be milled/printed.

Surgical procedure:

Routine site preparation regarding L.A injections and surgical site disinfections. A maxillary vestibular incision will be made from the maxillary second premolar on one side to the contralateral tooth. The incision will be made 5 mm above the mucogingival junction to leave an adequate cuff for closure. A full thickness mucoperiosteal flap will be reflected to expose the anterior and lateral maxillary walls. Superiorly the reflection exposes the pyriform rim, lateral nasal wall and the infraorbital nerve. Moving backwards, exposure of the zygomatico maxillary buttress is done followed by the maxillary tuberosity and finally the pterygomaxillary junction. The cutting guides will then be placed on the exposed maxilla. The cutting guides will have holes designed in them corresponding to the position of the fixation screws and a slot marking the level of the level of the Le fort 1 osteotomy which will be made using a reciprocating saw. The osteotomy is initiated and the cutting guide is removed.

The nasal septum, both lateral nasal walls and both pterygomaxillary junctions will be osteotomized using a mallet and a chisel and the maxilla finally down fractured and mobilized using Rowe's disimpaction forceps.

Without the use of inter maxillary fixation on an interocclusal wafer. the two-piece PSI will be placed and fixated above the level of the osteotomy using Mini screws. The mobile maxilla is moved until its one and only preplanned position is achieved using the PSI anatomical contours and then the maxilla is fixed. Copious irrigation is done and wound closure using an air cinch and a V-Y closure.

Post-Operative:

Immediate post-operative instructions and medications including analgesics and antibiotics will be given to the patient.

CT scan will be done 4 months post operatively. Then the preoperative and postoperative models will be superimposed to determine the accuracy of the surgically positioned maxilla, comparing it to the virtual plan.

• Control Group

The surgical procedure:

The exact same procedure will be repeated for the control group with the only difference being the fixation device which will consist of a one piece PSI spanning along the entire length of the osteotomy from one zygomaticomaxillary buttress to another.

Post-Operative:

Immediate post-operative instructions and medications including analgesics and antibiotics will be given to the patient.

CT scan will be done 4 months postoperatively.

Strategies to improve adherence to intervention protocols:

Assuring the accuracy of the patient specific fixation by printing skull models of the performed surgery and checking the plates. And such accuracy measures will be photographed and archived.

Criteria for discontinuing allocated interventions for a participant:

* Significant deviation from the virtual plan which will compromise the treatment outcome.
* Hardware failure (Non healing wound dehiscence, screw loosening, plate fracture, etc.)

Relevant concomitant care and interventions that are permitted:

- The application of postoperative elastics for minor occlusal adjustments. Relevant concomitant care that will be prohibited is the fixation of the separated maxilla in a position other than that dictated by the cutting and drilling guide

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with dentofacial deformity: skeletal class 2, class 3, vertical maxillary excess, Facial asymmetry.
* Patient seeking definitive surgical correction and refusing orthodontic camouflage.
* Maxillary impaction, advancement and rotations.
* Highly motivated patients.
* Good oral hygiene.
* Patients willing for the surgical procedure and follow-up, with an informed consent

Exclusion Criteria:

* Medically compromised patients
* Uncooperative patients
* Poor oral hygiene
* Periodontal diseases
* Patients with no desire for surgical correction
* Patients with any diseases that compromise bone or soft tissue healing Patients with local pathology that interfere with the bone healing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-05 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Stability of the new maxillary position | 4 months
  Primary outcome will be the positional stability of the repositioned maxilla which will be measured via CT scan by superimposing the postoperative maxillary segment obtained from a 4 months postoperative CT

SECONDARY OUTCOMES:
Intra-operative time | Intra-operative
  stop watch is used toc calculate the intra-operative time
Patient satisfaction using Visual Analogue Scale | 3 months
  Patient satisfaction will be gauged using VAS 3 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
Participants agreed to be part of the study but denied sharing any personal data